CLINICAL TRIAL: NCT04651725
Title: Effectiveness of Hippotherapy Simulator on Balance and Knee Strength in People With Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: Effectiveness of Hippotherapy Simulator in PwMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Ali Yavuz Karahan, Chairman of the Department of Rehabilitation Medicine, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Usak222
Record Dates: First submitted 2020-11-15; First posted 2020-12-03 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis; Exercise
Keywords: hippotherapy; multiple sclerosis; balance; strength; exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized pretest-posttest control group design
Who Masked: Outcomes Assessor
Masking Description: a blind physiotherapist will assess the study in outcomes in all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group 1: Exercise via mechanical horse-riding simulator (Active Comparator): All patients in both groups were planned to complete exercise sessions 3 times a week for 12 weeks, each lasting 35 minutes per day.
  Interventions: Other: Exercises
- Exercise group 2: Home exercises (Active Comparator): Home exercises will be consist of a warm-up, stretching, balance, back walking, fingertip walking exercises, the first of which is shown by the physiatrist or physiotherapist to the patients. These patients will be called twice a month to ask whether they have done the exercises, and the patients whose participation rate is below 80% will be excluded from the study by following the exercise schedule when they come to the physician's control monthly.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Patients were planned to complete exercise sessions 3 times a week for 12 weeks, each lasting 35 minutes per day.

SUMMARY:
A mechanical horse-riding simulator (MHRS) is a robotic device with a dynamic saddle that mimics the movement of a horse for purpose of hippotherapy. By simulating the rhythmic movements of the horse MHRS aims to increase the patient's balance, flexibility and adaptation and to provide postural adjustment. MHRS is supposed to produce walking patterns of a horse in a three-dimensional aspect. Movements in rhythmic repetitions improve postural coordination, allow to produce a reciprocal pattern. By simulating the rhythmic movements of a horse, MHRS aims to increase the patient's balance, flexibility and adaptation and to provide postural adjustment. This study aims to research the potential benefits of the mechanical horseback riding simulator on the postural balance and symptoms of multiple sclerosis patients.

DETAILED DESCRIPTION:
Hippotherapy or therapeutic horseback riding therapy is a form of animal-assisted therapy that uses the horse as a modality that aims to improve postural control, balance and mobility. With hippotherapy, it is aimed to change the center of gravity by using the movements of the horse and to ensure the adaptation of the trunk and pelvis by developing righting and balance reactions against this new position. Current studies suggest that hippotherapy may be a useful complementary treatment approach for improving balance, fatigue, spasticity, walking and quality of life in MS patients. However, horseback riding therapy itself has some limitations as a treatment due to costs, location and risks. By its nature horse-riding is too dynamic for patients and requires a large outdoor space.

This prospective clinical study aims to show potential benefits of horse riding in people with Multiple Sclerosis (PwMS) via a mechanical simulator.

Primer outcomes of the study are postural balance and muscle strength. Sample size calculation was performed and forty patients (inclusion and exclusion criteria will listed separately) were planned to be included in the study.

Participants will be allocated to the different treatment groups using the block randomization method.

All patients in both groups will planned to complete exercise sessions 3 times a week for 12 weeks, each lasting 35 minutes per day.

For the Group 1 (horse-riding simulator group), patients will will perform a horse riding simulation exercise at speeds of 15km/h, 18km/h, 20km/h, 22km/h, 25km/h, each lasting 5 minutes after warm-up for 5 minutes in each session. Then they will rest for 5 minutes.For the safety, a physiotherapist will be accompanied to the exercises for this group.

For the Group 2 (home exercise group) patients will perform home exercises. Home exercises will be consist of a warm-up, stretching, balance, back walking, fingertip walking exercises, the first of which is shown by the physiatrist or physiotherapist to the patients. These patients will be called twice a month to ask whether they have done the exercises, and the patients whose participation rate is below 80% will be excluded from the study by following the exercise schedule when they come to the physician's control monthly.

All participants will be filled with My Multiple Sclerosis (MMMS) scale, Berg Balance Scale (BBS), Timed Up and Go Test, before treatment and at the end of the 12th week. Quadriceps muscle strength will be measured with the microFET®2 Dynamometer before treatment and at the end of the 12th week.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient.
* Minimum age of 18 years
* Confirmed multiple sclerosis diagnosis.
* Expanded Disability Status Scale (EDSS) score below seven

Exclusion Criteria:

* Any vision or hearing problems,
* The presence of other neurological, orthopedic or rheumatic problems that may limit shoulder-pelvic movement or cause pain,
* Presence of physically disabled or uncontrolled chronic systemic disease,
* Having had a major trauma,
* To receive treatment for shoulder, hip, knee problems in the last 6 months,
* Having had an MS attack in the last 3 months.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Balance dysfunction in Multiple Sclerosis | At the end of the 12th week of exercise schedule
  The Balance will be measured with the "The Timed Up & Go (TUG)". TUG provides useful outcomes related to reduced falls risk.
  In patients with multiple sclerosis the Minimally Detectable Change was 3.5 seconds.
  Four teen seconds accepted as cut of scores (indicating risk of falls).
Muscle Strength | At the end of the 12th week of exercise schedule
  Quadriceps muscle strength will be measured with the microFET2 Dynamometer. The wireless microFET®2 Digital Handheld Dynamometer muscle tester is an accurate, portable Force Evaluation and Testing device. It is a modern adaptation of the time-tested art of hands-on manual muscle testing. Measurement Range 0-300 lbs force.

SECONDARY OUTCOMES:
Disability associated with Multiple Sclerosis | At the end of the 12th week of exercise schedule
  Disability associated with Multiple Sclerosis will be detected with The Expanded Disability Status Scale.
  The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a physiatrist.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Y Karahan, MD, Study Chair — University of Usak
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No